CLINICAL TRIAL: NCT07274267
Title: The Effect of Inspiratory Muscle Training on the Functional Status of Patients With Inflammatory Myopathy
Brief Title: Inspiratory Muscle Training in Patients With Inflammatory Myopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Józef Piłsudski University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: KB/91/2024
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Inflammatory Myopathies
Keywords: Inspiratory muscle training; Diaphragm ultrasound; Respiratory muscle strength; Exercise tolerance
MeSH Terms: conditions — Myositis

STUDY DESIGN:
Intervention Model Description: This is a single-group, prospective pilot intervention study evaluating the effects of inspiratory muscle training on functional status in patients with inflammatory myopathy. All participants receive the same inspiratory muscle training program and are followed for 12 months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inspiratory Muscle Training (IMT) (Experimental): Patients with inflammatory myopathy will perform a 3-month inspiratory muscle training (IMT) program using a threshold device (Philips Respironics Threshold IMT). Training will be home-based, preceded by individual instruction, and monitored through exercise diaries and follow-up phone consultations. Assessments will be performed before training, after 3 months, and during follow-up visits.
  Interventions: Behavioral: Inspiratory Muscle Training (IMT)

INTERVENTIONS:
Behavioral: Inspiratory Muscle Training (IMT) — Inspiratory muscle training performed with a threshold loading device (Threshold IMT, Philips Respironics). Participants perform 30 breaths once daily, 7 days per week, for 3 months. The training load is set at 30% of maximal inspiratory pressure (MIP) and increased by 10% if the perceived exertion decreases on two consecutive training days. Participants receive individualized instruction and regular follow-up consultations (every 2 weeks) to adjust load and verify adherence.

SUMMARY:
Inflammatory myopathies are rare autoimmune diseases leading to progressive muscle weakness, often including the respiratory muscles. This study aims to investigate whether inspiratory muscle training (IMT) using a threshold device can improve functional status in patients with inflammatory myopathy. Thirty-three patients will undergo a 3-month home-based IMT program with progressive resistance. Functional capacity, inspiratory muscle strength, lung function, diaphragmatic mobility, fatigue, and quality of life will be assessed at baseline and during follow-up. The primary hypothesis is that IMT will enhance inspiratory muscle strength and translate into better functional performance and quality of life.

DETAILED DESCRIPTION:
Idiopathic inflammatory myopathies (IIM) are rare autoimmune disorders characterized by progressive, symmetrical proximal muscle weakness, frequently affecting the respiratory muscles. Diaphragmatic dysfunction and reduced inspiratory muscle strength contribute to impaired ventilation, fatigue, and reduced exercise tolerance. While exercise training has proven beneficial in patients with various neuromuscular conditions, evidence regarding inspiratory muscle training (IMT) in IIM is lacking.

This pilot interventional study will prospectively evaluate the impact of a 3-month IMT program on respiratory and functional outcomes in patients with IIM. The intervention consists of daily inspiratory resistance training (30 breaths/day, 7 days/week) using the Threshold IMT device (Philips Respironics, USA). Training intensity is set at 30% of maximal inspiratory pressure (MIP) and adjusted progressively based on patient-reported exertion. Participants receive individualized instruction, follow-up phone consultations every 2 weeks, and record adherence in exercise diaries.

Assessments include inspiratory muscle strength (MIP measured with Powerbreathe KH2 and RP Check), spirometry (FEV1, FVC, FIVC, IRV), diaphragm ultrasound (mobility and thickness fraction), six-minute walk test (6MWT), fatigue assessment (Borg scale, Fatigue Severity Scale), and quality of life (SF-36). Outcomes will be measured 3 months before training, at baseline, after 3 months of training, and during extended follow-up (up to 6-12 months). The primary endpoint is change in MIP. Secondary endpoints include pulmonary function parameters, diaphragmatic function, exercise tolerance, fatigue, and health-related quality of life.

The study will be conducted in the Neurology Clinic of the Medical University of Warsaw (WUM). A total of 33 patients with IIM, diagnosed according to EULAR/ACR criteria, will be recruited. Inclusion requires age ≥18 and written informed consent. Exclusion criteria include cognitive impairment, acute respiratory infection, prior respiratory training, pneumothorax, pulmonary hypertension, or contraindications to IMT. This trial is expected to provide the first structured evidence on the role of IMT in improving functional status in patients with inflammatory myopathy, potentially guiding individualized rehabilitation strategies for this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of inflammatory myopathy according to EULAR/ACR criteria
* Age ≥ 18 years
* Stable clinical condition allowing participation in physical activity
* Ability to understand and follow instructions
* Written informed consent to participate in the study

Exclusion Criteria:

* Cognitive impairment preventing proper exercise performance
* Current respiratory tract infection
* Previous respiratory muscle training within the last 12 months
* History of spontaneous pneumothorax
* Pulmonary hypertension
* Tympanic membrane rupture or other middle ear pathology
* Lack of voluntary and informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in maximal inspiratory pressure (MIP) | 3 months before training, baseline, 3 months (end of training), 6 months, 9 months, 12 months
  Maximal inspiratory pressure measured at the mouth using Powerbreathe KH2 and RP Check devices. MIP reflects inspiratory muscle strength and is expressed in cmH₂O.

SECONDARY OUTCOMES:
Change in forced vital capacity (FVC) | 3 months before training, baseline, 3 months (end of training), 6 months, 9 months, 12 months
  Spirometric measurement of forced vital capacity performed using the NDD EasyOne device. Results expressed as absolute and percent predicted values.
Change in forced expiratory volume in 1 second (FEV1) | 3 months before training, baseline, 3 months (end of training), 6 months, 9 months, 12 months
  Spirometric assessment of airway function, expressed as FEV₁ (L and % predicted).
Change in diaphragm thickness | 3 months before training, baseline, 3 months (end of training), 6 months, 9 months, 12 months
  Ultrasound assessment of diaphragm thickening fraction using Philips Lumify linear probe.
Change in 6-Minute Walk Distance (6MWD) | 3 months before training, baseline, 3 months (end of training), 6 months, 9 months, 12 months
  Functional exercise capacity assessed by the 6-Minute Walk Test (6MWT), conducted on a 25 m corridor. Distance covered in 6 minutes is recorded in meters.
Change in perceived exertion (Borg Scale) | 3 months before training, baseline, 3 months (end of training), 6 months, 9 months, 12 months
  Subjective fatigue during exertion assessed using the modified Borg Rating of Perceived Exertion (0-10).
Change in fatigue severity (Fatigue Severity Scale) | 3 months before training, baseline, 3 months (end of training), 6 months, 9 months, 12 months
  Assessment of perceived fatigue using the Fatigue Severity Scale (FSS).
Change in quality of life (SF-36) | 3 months before training, baseline, 3 months (end of training), 6 months, 9 months, 12 months
  Assessment of health-related quality of life using the 36-Item Short Form Health Survey (SF-36), including physical and mental health domains.

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinical Center of the Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study involves a small sample of clinical patients and contains potentially identifiable medical information. Summary results will be made available through scientific publications and presentations.

REFERENCES:
- [Background] Van Thillo A, Vulsteke JB, Van Assche D, Verschueren P, De Langhe E. Physical therapy in adult inflammatory myopathy patients: a systematic review. Clin Rheumatol. 2019 Aug;38(8):2039-2051. doi: 10.1007/s10067-019-04571-9. Epub 2019 May 21. PMID 31115788
- [Background] Ashton C, Paramalingam S, Stevenson B, Brusch A, Needham M. Idiopathic inflammatory myopathies: a review. Intern Med J. 2021 Jun;51(6):845-852. doi: 10.1111/imj.15358. PMID 34155760
- [Background] Lundberg IE, Miller FW, Tjarnlund A, Bottai M. Diagnosis and classification of idiopathic inflammatory myopathies. J Intern Med. 2016 Jul;280(1):39-51. doi: 10.1111/joim.12524. PMID 27320359
- See also: Academy of Physical Education in Warsaw - institutional website — https://www.awf.edu.pl/en